CLINICAL TRIAL: NCT01891084
Title: A Randomized Controlled Trial on the Effect of Fever Suppression by Antipyretics on Influenza
Brief Title: The Benefit and Harm of Fever Suppression by Antipyretics in Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Dennis Kai-Ming Ip, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKMI003.4
Record Dates: First submitted 2013-06-19; First posted 2013-07-02 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Influenza
Keywords: Influenza; Antipyretics; Fever
MeSH Terms: conditions — Influenza, Human; Fever | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Paracetamol 1 tablet (500mg) four times daily. For a maximum period of 5 days if the patient is still having fever. When required, participants may take up to 2 tablets (1gm) in each dose. Precautionary statement (Do not exceed 8 tablets daily) will be printed on the dispensary label to avoid overdose.
  Backup NSAID ibuprofen 200mg orally every 8 hourly will also be provided to all participants, which can be taken when necessary (PRN) if the participant finds the fever intolerable.
  Interventions: Drug: Paracetamol; Drug: Backup NSAID ibuprofen
- Placebo (Placebo Comparator): (Identical-looking) Placebo 1 tablet four times daily. For a maximum period of 5 days if the patient is still having fever. When required, participants may take up to 2 tablets in each dose. Precautionary statement (Do not exceed 8 tablets daily) will be printed on the dispensary label to avoid overdose.
  Backup NSAID ibuprofen 200mg orally every 8 hourly will also be provided to all participants, which can be taken when necessary (PRN) if the participant finds the fever intolerable
  Interventions: Drug: Placebo; Drug: Backup NSAID ibuprofen

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 1 tablet (500mg) four times daily. For a maximum period of 5 days if the patient is still having fever. When required, participants may take up to 2 tablets (1gm) in each dose.
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Placebo — (Identical-looking) Placebo 1 tablet four times daily. For a maximum period of 5 days if the patient is still having fever. When required, participants may take up to 2 tablets in each dose.
  Arms: Placebo
Drug: Backup NSAID ibuprofen — Backup NSAID ibuprofen 200mg orally every 8 hourly will also be provided to all participants, which can be taken when necessary (PRN) if the participant finds the fever intolerable.
  Other Names: ibuprofen

SUMMARY:
The purpose of this study is to investigate the potential benefits and risks of antipyretics use in naturally occurring influenza virus infections in humans.

DETAILED DESCRIPTION:
Background:

Being one of the commonest conditions encountered in modern medical practice, fever is commonly regarded as an illness that has to be treated, both by medical professionals and patients. However, objective and convincing evidence is lacking that naturally occurring fever is harmful, and there is growing evidence that fever may serve an important host defense mechanism in infections and the risks of its suppression may far outweigh its apparent benefits. In acute respiratory infections including influenza, antipyretics are commonly being prescribed as a symptomatic treatment. Evidence from different randomized controlled trials, however, had challenged the actual amount of clinical benefit achievable by fever suppression for improving the patients' comfort and behavior. On the other hand, evidence from animal and human challenge studies has suggested that antipyretic therapy may actually prolong the duration of illness, suppress humoral antibody response, and increase the level and duration of viral shedding.

The knowledge gap:

Most of the currently available evidence on the harms and benefits of antipyretic treatment of upper respiratory tract infections (URTIs) are from either experimental animal studies, or human challenge studies with various respiratory viruses, or from randomized controlled trials (RCTs) on patients with fever of presumed viral origin. There has yet been no RCT that has investigated on the effect of antipyretics on the clinical course, disease duration, and the pattern of viral shedding in naturally occurring acute URTIs of viral origin in humans. Whereas acute URTIs can be caused by a range of viral and non-viral causes, influenza virus infection is one of its leading cause, and its pathogenesis is relatively well understood compared to some other respiratory viruses.

Aim:

To investigate the potential benefits and risks of antipyretic use in naturally occurring influenza virus infections in humans.

Design and subjects:

The study is a double-blind, randomized controlled trial. Four hundred young adults aged 18-30 years will be recruited when they present with symptoms of acute respiratory infection within 48 hours of symptoms onset to university health clinics, and being tested positive with a QuickVue rapid influenza test. They will receive their clinical consultation and prescriptions as indicated as usual, and being randomized to receive either paracetamol or placebo, and given back-up NSAID for intolerable fever when required. Blood specimen, nasal and throat swabs will be collected on the same day (day 1). They will be followed-up on day 4, day 7 and day 10 for further collection of nasal and throat swabs, and on day 28 for a final blood taking. A symptom diary will be kept by each participant for 10 days for monitoring the clinical course of the infection.

Potential significance:

This will be the first RCT to investigate the effect of antipyretics on the clinical course, disease duration, and the pattern of viral shedding in naturally occurring influenza virus infection in humans. Findings from this study will have important contribution to our understanding on the role of fever as a host defense mechanism, and help to inform the appropriate clinical management approach in human influenza virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-30
* Presenting with symptoms of acute URTI (at least two among the following symptoms: body temperature ≥37.8°C, cough, rhinorrhea, sore throat, headache, myalgia/arthralgia) within 48 hours of illness onset
* being tested positive with a QuickVue rapid influenza test

Exclusion Criteria:

* Allergic to paracetamol or any other antipyretics
* Have any underlying immunocompromized condition or be receiving immunosuppressive agents.
* Have any history of chronic liver disease, or any active lung, heart or renal diseases requiring regular medication.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time from recruitment to illness resolution, defined as the time when fever and at least nine out of the ten influenza symptoms had subsided (graded as 0 by the patient) for a period of 24 hours. | 10 days
  Self-recording of temperature twice daily for ten days (D1-D10) will be performed and recorded using a standard tympanic thermometer provided for free to each participant. Participants will also keep symptom diary twice daily for 10 days (from D1-D10), using 4-point scale of 0, 1, 2, or 3 for absent, mild, moderate, or severe symptoms respectively. Mild symptoms are easily tolerated and do not interfere with any usual activities; moderate symptoms interfere with usual activities; Severe symptoms are such that the individual cannot carry out usual activities. Ten common influenza symptoms (including feverishness, chills, cough, rhinorrhea, sore throat, general fatigue, headache, myalgia/arthralgia, vomiting, and diarrhea) will be recorded.
Time from recruitment to cessation of viral shedding, defined as the time when no virus is detected by RT-PCR from both nasal and throat swabs. | 10 days
  Nasal and throat swabs will be collected on D1, D4, D7 and D10 for viral identification and subtyping by viral culture, and viral load detection and quantification by quantitative RT-PCR.

SECONDARY OUTCOMES:
Time to cessation of illness and viral shedding from illness onset | 10 days
  Nasal and throat swabs will be collected on D1, D4, D7 and D10 for viral identification and subtyping by viral culture, and viral load detection and quantification by quantitative RT-PCR.
The duration of individual symptoms | 10 days
  Participants will keep symptom diary twice daily for 10 days (from D1-D10), using 4-point scale of 0, 1, 2, or 3 for absent, mild, moderate, or severe symptoms respectively. Mild symptoms are easily tolerated and do not interfere with any usual activities; moderate symptoms interfere with usual activities; Severe symptoms are such that the individual cannot carry out usual activities. Ten common influenza symptoms (including feverishness, chills, cough, rhinorrhea, sore throat, general fatigue, headache, myalgia/arthralgia, vomiting, and diarrhea) will be recorded for ten days (D1-D10) and the duration of individual symptoms will be assessed.
The incidence of secondary complications | 10 days
  The symptom diary will be checked on each follow-up (D4, D7, and D10) and collected on D10 by our research staff when the patient returns for follow-up. Symptoms of possible side effects related to treatment (including skin rashes, nausea, vomiting, jaundice, dark urine) will be recorded. The occurrence of any complications including otitis media, bronchitis, sinusitis, and pneumonia will be enquired during all follow-up sessions and recorded, and cross checking with the attending doctor will be done where necessary.
The use of backup NSAID provided | 10 days
  Compliance on the trial medication (paracetamol/ placebo) and the use of the backup NSAID prescribed on a PRN basis will also be recorded in the symptom diary.
Quality of life | 10 days
  A simple quality of life (QOL) assessment based on two simple validated 11- point visual analog scales will also be done daily by all participants form D1 - D10, one to rate their own ability for performing normal daily activities (0 = unable to perform normal activity to 10 = fully able to perform normal activity) , and the other for a self-perceived overall health status over a 24-hour (0 = worst health to 10 = best possible health), both of which will be compared to an initial assessment of their normal pre-influenza state reported on the D1 baseline. All participants will also be required to complete the Acute Form of the Short Form-36, version 2 (SF-36), in D1, D10 and D28, for a more details assessment on the changes of Health-related quality of life (HRQL) related to the episode of the influenza infection.
Geometric mean rise in antibody titre against the infecting type or subtype of influenza virus | 28 days
  Paired sera will be collected on D1 and D28 for measuring the humoral antibody titres against the infecting type or subtype and other circulating strains of influenza viruses, and for evaluating the geometric mean titer rise from baseline to convalescence.
The severity of individual symptoms | 10 days
  Participants will keep symptom diary twice daily for 10 days (from D1-D10), using 4-point scale of 0, 1, 2, or 3 for absent, mild, moderate, or severe symptoms respectively. Mild symptoms are easily tolerated and do not interfere with any usual activities; moderate symptoms interfere with usual activities; Severe symptoms are such that the individual cannot carry out usual activities. Ten common influenza symptoms (including feverishness, chills, cough, rhinorrhea, sore throat, general fatigue, headache, myalgia/arthralgia, vomiting, and diarrhea) will be recorded for ten days (D1-D10) and the severity of individual symptoms will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis KM Ip, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- University Health Service, The Hong Kong Polytechnic University, Hong Kong, Hksar, China